CLINICAL TRIAL: NCT03478852
Title: Investigating Epilepsy: Screening and Evaluation
Status: Recruiting | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 180066; 18-N-0066
Record Dates: First submitted 2018-03-15; First posted 2018-03-27 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10-24

CONDITIONS: Seizures; Epilepsy; Epilepsy, Temporal Lobe; Partial Epilepsy
Keywords: Seizure Disorder; Seizures; Antiepileptic Drug; Natural History Study; Screening Protocol
MeSH Terms: conditions — Seizures; Epilepsy; Epilepsy, Temporal Lobe; Epilepsies, Partial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Arm: Single arm open enrollment of patients with standard of care treatment and evaluation

SUMMARY:
Background:

Epilepsy affects about 1 percent of the U.S. population. Most people with epilepsy respond well to medicine, but some do not. Researchers want people who have diagnosed or suspected epilepsy to participate in ongoing studies. They want to learn more about clinical care for epilepsy. They want fellows and residents to learn more about the care of people with epilepsy.

Objectives:

To learn more about seizures and find ways to best treat people with drug-resistant epilepsy.

Eligibility:

Adults and children ages 8 years and older with diagnosed or suspected epilepsy

Design:

Participants will be screened with:

Physical exam

Medical history

Questionnaires

Participants will have many visits. They may be admitted to the hospital for several weeks. Their medication might be stopped or changed.

Participants will have many tests:

Blood and urine tests

EEG: Wires attached to the head with paste record brain waves. This may be videotaped.

Thinking and memory tests

MRI: Participants lie on a table that slides in and out of a tube. They perform simple tasks in the tube.

MEG: Participants lie on a table and place their head in a helmet to record brain waves.

PET scan: Participants lie on a table that slides into a machine. A small amount of radioactive dye is injected into their arm with an IV. For the IV, a small tube is inserted into the arm with a needle.

Participants will stay enrolled in this study if they join other epilepsy-related studies. They may be contacted at intervals for follow-up. Their participation will end if they have not been seen clinically for their epilepsy for 3 years.

DETAILED DESCRIPTION:
Study Description:<TAB>

This protocol is designed to serve as a screening protocol that provides standard evaluation and treatment for patients with epilepsy. Clinical data collected through this protocol will be used in other NIH epilepsy-related research to screen for eligibility in the respective protocols and may also be used for descriptive and/or correlative research through this protocol.

Objectives:

Primary Objective:

Maintain a cohort of patients who are referred to the NIH with a known or suspected diagnosis of epilepsy that can be accessed by other NIH studies to screen for eligibility to participate in ongoing epilepsy-related protocols.

Secondary Objectives:

* to follow the natural history of subjects with epilepsy and epilepsy and related disorders, and
* to allow for descriptive and/or correlational studies based on the data collected through clinical care of these patients.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 8 years or older
* Known or suspected diagnosis of epilepsy
* Ability to give informed consent or have a legally authorized representative able to give consent (for adults without consent capacity) or parent/guardian able to provide informed consent (for a child)
* If unable to give informed consent, ability to give assent (for minors 8 and older)

EXCLUSION CRITERIA:

* Patients with unstable medical conditions that, in the opinion of the investigators, makes participation unsafe, or who, in the opinion of the investigators may be unable to comply with the protocol
* Patients who are unable to travel to the NIH

Ages: 8 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults and Children age 8 years and older referred with a known or suspected diagnosis of epilepsy
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-03-28 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Screening and characterization of patients with drug-resistant epilepsy for epilepsy-related protocols | 5 year period
  to characterization of patients epilepsy to determine their eligibility for inclusion in other epilepsy-related protocols.

SECONDARY OUTCOMES:
Data obtained through clinical care will provide descriptive and/or correlative research | 5 year period
  data obtained through clinical care provided under this protocol in descriptive and/or correlative research in this and other protocols.

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Tajali, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2018-N-0066.html